CLINICAL TRIAL: NCT07351981
Title: Randomized Double-Blind Study to Evaluate the Efficacy of Transcutaneous Pulsed Radiofrequency (PRF) Treatment for Knee Pain
Brief Title: TcPRF for Knee Osteoarthritis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Martina Rekatsina, Assisitant Professor Of Anaesthesiology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 695/24-07-2025
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Knee OA; Knee Osteoarthristis
Keywords: knee; osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: * Type: Randomized, double-blind, sham-controlled study.
  * Duration: 6 months
  * Study Population: Adults aged 40-75 years with chronic knee pain (lasting ≥ 6 months) due to osteoarthritis (OA).
  * How many patients in each group: 25 patients in each group (according to Janssens et al, 2024)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind, assessor masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TcPRF (Active Comparator): Transcutaneous pulsed RF -connected to treatment mode of the spring pulsed rf generator
  Interventions: Device: Transcutaneous Pulsed Radiofrequency (PRF) Treatment for Knee Pain
- TcPRF sham (Sham Comparator): sham of transcutaneus pRF- connected to demo mode of the spring pulsed rf generator
  Interventions: Device: sham treatment of pulsed rf on knee

INTERVENTIONS:
Device: Transcutaneous Pulsed Radiofrequency (PRF) Treatment for Knee Pain — application of TcPRF patches
  Arms: TcPRF
Device: sham treatment of pulsed rf on knee — Transdermal patch will be connected to demo mode of the spring pulsed rf generator. no treatment will be given
  Arms: TcPRF sham

SUMMARY:
Objectives

* Primary Objective: To evaluate the efficacy of transcutaneous PRF treatment in reducing knee pain compared to a sham intervention
* Secondary Objectives: To assess the improvement in functional outcomes and patient satisfaction following PRF treatment.

Study Design

* Type: Randomized, double-blind, sham-controlled study.
* Duration: 6 months
* Study Population: Adults aged 40-75 years with chronic knee pain (lasting ≥ 6 months) due to osteoarthritis (OA).
* How many patients in each group: 25 patients in each group (according to Janssens et al, 2024) Inclusion Criteria
* Diagnosed with knee osteoarthritis according to NICE criteria.
* Chronic knee pain (Visual Analogue Scale [VAS] ≥ 4).
* Failure to respond adequately to conventional treatments (e.g., NSAIDs, physical therapy).
* Willingness to comply with study procedures. Exclusion Criteria
* Previous PRF/RF treatment for knee pain.
* Hyaluronic acid injection for knee pain in the past 6 months
* Knee surgery within the last 6 months.
* Severe cardiovascular, neurological, or psychiatric conditions.
* Active systemic infections or local skin infections at the knee.
* Pregnancy or lactation.

DETAILED DESCRIPTION:
Randomization and Blinding

* Randomization: Participants will be randomly assigned to one of two groups: PRF treatment or sham.
* Blinding: Both participants and investigators will be blinded to the treatment allocation. The device used for PRF treatment will have an identical appearance for both the active and sham groups, but the sham electrode will not deliver active treatment.

Intervention Both groups will receive disposable electrodes on either side of the knee: one skin electrode on the inside and one on the outside of the knee.

* PRF Group: Participants will receive PRF treatment using a specific protocol (e.g., 3 Hz, 5 ms, 15 minutes, 3 sessions with 1 week and 3 weeks interval). The output will be adjusted according to the distance between electrodes in cm. This will be between 0.7A (circumference 23cm) and 1.4A for 38cm (Spring 2, Clinical Guidelines, Table 1)
* Sham Group: Participants will receive a sham treatment using a device identical in appearance but without delivering the actual PRF therapy.

Outcome Measures Primary Outcome • Pain Reduction: Measured using the NRS (numerical rating scale) at baseline, immediately after treatment, and at follow-up intervals (2 weeks, 4 weeks, 8 weeks, 12 weeks).

Secondary Outcomes

* Functional Improvement: Assessed using the Western Ontario and McMaster Universities Arthritis Index (WOMAC) scores.
* Patient Satisfaction: Measured using a Likert scale for overall satisfaction with treatment.
* Global Assessment: Patient's global assessment of change in pain and function.
* Medication reduction Sample Size Calculation
* Estimate: Based on previous studies and expected effect size, calculate the necessary sample size to achieve a power of 80% and a significance level of 0.05. The sample size must account for potential dropouts.

Data Collection and Management

* Data will be collected at baseline, post-treatment, and during follow-up visits.
* Use electronic case report forms (eCRFs) for data entry.
* Ensure the security and confidentiality of participant data. Statistical Analysis
* Primary Analysis: Compare the mean change in VAS scores between the PRF and sham groups using an independent t-test or ANCOVA, adjusting for baseline values.
* Secondary Analysis: Compare changes in WOMAC scores and patient satisfaction between groups using similar statistical methods.
* Responder Analysis: Define responders as those with ≥30% reduction in VAS scores from baseline and compare proportions between groups using a chi-square test.
* Intention-to-Treat (ITT) Analysis: Include all randomized participants in the analysis based on the treatment they were allocated, regardless of whether they completed the study.

Ethical Considerations

* Obtain informed consent from all participants.
* Ethical approval from a recognized Institutional Review Board (IRB) is required.
* Ensure that participants can withdraw at any time without affecting their standard care.

Monitoring and Safety

* Adverse Events: Monitor and record all adverse events during the study.
* Data Safety Monitoring Board (DSMB): Establish a DSMB to review safety data periodically.

Dissemination of Results

• Results will be published in a peer-reviewed journal and presented at relevant conferences within a year after results are known. Data will be reported according to CONSORT guidelines.

Timeline

* Recruitment Period: 3 months
* Intervention Period: 4 weeks
* Follow-up Period: 3 and 6 months
* Data Analysis and Reporting: 3 months after study completion.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with knee osteoarthritis according to NICE criteria.
* Chronic knee pain (Visual Analogue Scale [VAS] ≥ 4).
* Failure to respond adequately to conventional treatments (e.g., NSAIDs, physical therapy).
* Willingness to comply with study procedures. Exclusion Criteria
* Previous PRF/RF treatment for knee pain.
* Hyaluronic acid injection for knee pain in the past 6 months
* Knee surgery within the last 6 months.
* Severe cardiovascular, neurological, or psychiatric conditions.
* Active systemic infections or local skin infections at the knee.
* Pregnancy or lactation.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction | 12 weeks
  Measured using the NRS (numerical rating scale) at baseline, immediately after treatment, and at follow-up intervals (2 weeks, 4 weeks, 8 weeks, 12 weeks).

SECONDARY OUTCOMES:
Functional Improvement | 12 weeks
  Assessed using the Western Ontario and McMaster Universities Arthritis Index (WOMAC) scores.
• Patient Satisfaction | 12 weeks
  Measured using a Likert scale for overall satisfaction with treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Aretaieion University Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided